CLINICAL TRIAL: NCT01573897
Title: Influence of Sleep Apnea Syndrome and Its Treatment by Positive Airway Pressure Therapy on Transcutaneous Oxygen Tension (PtcO2) in Patients With Foot Wound or at Risk for Foot Wound
Brief Title: Impact of Sleep Apnea on Diabetic Foot Wound.
Acronym: SAS-FOOT
Status: Terminated | Type: Observational
Why Stopped: Difficulty including subjects corresponding to the criteria.
Sponsor: AGIR à Dom (Other)
Responsible Party: Sponsor
Other Study IDs: 12-AGIR-01
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Foot; Sleep Apnea
Keywords: Diabetes; Sleep apnea; Diabetic foot; Microcirculation
MeSH Terms: conditions — Diabetic Foot; Sleep Apnea Syndromes; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Foot-wound without SAS: patients with diabetic foot wound(or at risk of diabetic foot wound) without sleep apnea syndrome
- Foot-wound with SAS: patients with diabetic foot wound(or at risk of diabetic foot wound) with sleep apnea syndrome

SUMMARY:
Sleep apnea syndrome (SAS) is a common comorbidity of type 1 and type 2 diabetes. A low transcutaneous oxygen tension (PtcO2) measured on the foot is pejorative prognostic factor for the healing of a diabetic foot wound. SAS causes intermittent nocturnal hypoxia and sympathetic overactivity. The investigators hypothesized that SAS could be a factor reducing the PtcO2.Therefore, the main objective of this study is to assess the variation in PtcO2 between the end of the night and midday in patients with -or at risk of- diabetic foot wound according to the presence or not of sleep apnea syndrome.The secondary objective is to address the microvascularisation of diabetic patients having foot wounds according to their status regarding sleep apnea syndrome.

DETAILED DESCRIPTION:
The study is observational, cross-sectional. Presence of sleep apnea syndrome will be assessed on the same night than the main outcome, that is the difference in PtcO2 between 5:00 AM and 12:00AM. Microvascularisation will be assessed by Laser Speckle Contrast Imaging Analysis (LASCA).

Sample size is estimated at 60 patients based on previous revascularisation studies having PtcO2 as main outcome.

An intermediary analysis is planned after 40 inclusions.

ELIGIBILITY:
Inclusion Criteria:

* Types 1 or 2 or MODY diabetes with diabetic foot wound (or at risk of foot wound stage 2 and 3 (see reference PMID:18442189).
* Patients covered by social insurance

Exclusion Criteria:

* Patients with sleep apnea syndrome previously treated by positive airway pressure therapy.
* Patients previously treated by additional oxygen therapy. Patient with unstable psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutives diabetic patients referred to our tertiary diabetes unit (Grenoble University Hopsital, France) for diabetic foot wound
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-06-04 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Transcutaneous oxygen tension (PtcO2) | Transcutaneous oxygen tension is assessed at the end of the night (5:00a.m) and at midday (12:00 a.m)
  Transcutaneous oxygen tension (PtcO2)is measured with a Radiometer TCM4 (Radiometer, Copenhagen, Denmark) device, on the dorsum of the foot at the base of the second metatarsal, or as close to this location as possible. Calibration is performed before each measurement. All measurements are performed in supine position after 20 min of rest. Room temperature is kept constant (around 21°C-24°C). Patients are asked to avoid smoking or drinking coffee for at least 2 h before investigations

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Borel, Pr MD PhD, Principal Investigator — Diabetes and Endocrinology Unit, Grenoble University Hospital
Locations (1):
- Diabetes and Endocrinology Unit, Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided